CLINICAL TRIAL: NCT05029999
Title: Phase 1 Pilot Study With Dose Expansion of Chemotherapy in Combination With CD40 Agonist and Flt3 Ligand in Metastatic HER2 Negative Breast Cancer
Brief Title: CD40 Agonist, Flt3 Ligand, and Chemotherapy in HER2 Negative Breast Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Celldex Therapeutics (Industry); Gateway for Cancer Research (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Sangeetha Reddy, Assistant Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCCC-03121; STU-2021-0657
Record Dates: First submitted 2021-08-25; First posted 2021-09-01 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: HER2-negative Breast Cancer; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — liposomal doxorubicin; flt3 ligand protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort A (Experimental): PLD chemotherapy will be administered 40 mg/m2 as intravenous injection once per cycle until toxicity or progression.
  CDX-1140 will be administered 1.5mg/kg as intravenous injection once per cycle until toxicity or progression for up to 24 months.
  CDX-301 will be administered 75µg/kg as subcutaneous injection daily x 5 days cycles 1 and 2 only.
  Interventions: Drug: PLD Chemotherapy; Drug: CDX-1140; Drug: CDX-301
- Cohort C (Experimental): PLD chemotherapy will be administered 40 mg/m2 as intravenous injection once per cycle until toxicity or progression.
  CDX-1140 will be administered 1.5mg/kg as intravenous injection once per cycle starting on cycle 2 until toxicity or progression for up to 24 months.
  CDX-301 will be administered 75µg/kg as subcutaneous injection daily x 5 days cycles 2 and 3 only.
  Interventions: Drug: PLD Chemotherapy; Drug: CDX-1140; Drug: CDX-301

INTERVENTIONS:
Drug: PLD Chemotherapy — PLD chemotherapy will be administered 40 mg/m2 as intravenous injection once per cycle.
  Other Names: Pegylated liposomal doxorubicin
Drug: CDX-1140 — CDX-1140 will be administered 1.5mg/kg as intravenous injection once per cycle.
  Other Names: CD40 monoclonal antibody
Drug: CDX-301 — CDX-301 will be administered 75µg/kg as subcutaneous injection daily x 5 doses per cycle for 2 cycles.
  Other Names: Flt3 Ligand

SUMMARY:
This research study is being done to find out if the immunotherapy drugs called CDX-301 and CDX-1140 in combination with the standard chemotherapy treatment pegylated liposomal doxorubicin (PLD, Doxil) are safe and effective at controlling the cancer in patients with metastatic triple Human Epidermal Growth Factor Receptor 2 (HER2) negative breast cancer, and to determine a safe dose and treatment schedule of the three drugs. This research study will also test how your immune system responds to these treatments alone and in combination.

DETAILED DESCRIPTION:
The immunotherapy drugs CDX-301 and CDX-1140 in combination with the standard chemotherapy treatment PLD work by kickstarting the immune response against cancer cells. CDX-301 increases the antigen presenting immune cells needed to kickstart the immune response, CDX-1140 activates these cells, and chemotherapy helps release antigens from the cancer cells to train these antigen presenting immune cells to recognize the cancer for the immune system to attack it.

Metastatic or unresectable triple negative breast cancer patients will receive this triplet combination that has been shown in preclinical studies to be more effective than the individual treatments or doublet combinations. To understand how the immunotherapies are working, some patients will receive the immunotherapy or chemotherapy only for one cycle prior to receiving the full triplet combination therapy. Ultimately, all patients will receive the triplet combination to study safety and how effective this treatment is at controlling triple negative breast cancer and improving survival outcomes.

The original design of the project includes 3 cohorts (arms). In February 2024 Cohort B (experimental arm) was closed to further enrollment.

Cohort B includes the following design:

PLD chemotherapy will be administered 40 mg/m2 as intravenous injection once per cycle starting on cycle 2 until toxicity or progression.

CDX-1140 will be administered 1.5mg/kg as intravenous injection once per cycle until toxicity or progression for up to 24 months.

CDX-301 will be administered 75µg/kg as subcutaneous injection daily x 5 days cycles 1 and 2 only.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable Stage III or Stage IV HER2 negative breast cancer (either triple negative or hormone receptor positive)

  * Triple negative breast cancer for this study is defined as estrogen receptor <10%, progesterone receptor <10% by immunohistochemistry, and HER2- negative by Herceptest (0 or 1+) or not amplified by in situ hybridization as per routine clinical testing.
  * Hormone receptor positive breast cancer for this study is defined as either estrogen receptor ≥10% or progesterone receptor ≥10% by immunohistochemistry, and HER2- negative by Herceptest (0 or 1+) or not amplified by in situ hybridization as per routine clinical testing.
* Age 18 years or older
* Performance status ECOG 0-2
* Life expectancy ≥ 12 weeks
* Documented progressive disease, based on radiographic, clinical or pathologic assessment, during or subsequent to last anticancer therapy. Patients who need to change systemic therapy for other indications such as toxicity that are otherwise eligible for this study may enroll with approval of the lead principal investigator.
* For triple negative breast cancer patients, subject is in first to fourth line setting of treatment for metastatic or unresectable disease, and have received 0 to 3 prior regimens for metastatic or unresectable disease.
* For hormone receptor positive breast cancer patients, subjects must have received prior cyclin dependent kinase inhibitor in the metastatic setting. They may have received up to 3 prior lines of chemotherapy and/or antibody drug conjugates for metastatic or unresectable disease.
* Among triple negative breast cancer patients enrolled in the first line treatment setting, subjects must be PD-L1 negative by 22C3 assay and not be eligible for FDA approved standard of care chemotherapy and anti-PD-1/PD-L1 combination therapy as alternative to this clinical trial. This does not apply if patients have previously received PD-1 or PD-L1 blockade as part of neoadjuvant or adjuvant therapy regimen.
* Screening laboratory values must meet the following criteria:

  * Neutrophils ≥ 1500/uL
  * Platelets ≥ 100 x10(9)/L
  * Hemoglobin ≥ 8 g/dL Patients may receive erythrocyte transfusions to achieve this hemoglobin level at the discretion of the investigator. Initial treatment must not begin earlier than the day after the erythrocyte transfusion.
  * Creatinine ≤ 2 mg/dL
  * Creatinine clearance >30 mL/minute
  * AST ≤ 2.5 X ULN without, and ≤ 5 x ULN with hepatic metastasis
  * ALT ≤ 2.5 X ULN without, and ≤ 5 x ULN with hepatic metastasis
  * Total Bilirubin ≤ 1.5 X ULN (except patients with Gilbert's syndrome or liver involvement, who must have a total bilirubin ≤ 2 X ULN)
  * Alkaline phosphatase ≤ 2.5 X ULN without, and ≤ 5 x ULN with hepatic metastasis
* All men as well as women of child bearing potential enrolled in this trial must agree to use effective contraception during the course of the trial and for at least 6 months after discontinuing study treatment. Patients and/or partners who are surgically sterile or postmenopausal are exempt from this requirement.

  * A female of child-bearing potential is any woman (regardless of sexual orientation, marital status, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria: ( 1) has not undergone a hysterectomy or bilateral oophorectomy OR (2) has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
* Provision of consent for pre-treatment and on-treatment biopsies. Biopsy sites must be soft tissue tumor lesions or accessible visceral diseases that can be biopsied with acceptable clinical risk (as judged by the investigator); are large enough to allow for the collection of tumor tissue for proposed correlative studies (e.g., anticipated goal of 6-8 cores preferred when feasible using a ≥ 18 gauge needle with an expected core sample length of 5 mm); and have not been irradiated prior to entry. This does not include bone lesions. This may exclude many lung lesions and small lesions.
* Measurable disease allowing for serial assessment of at least one target lesion(s) by RECIST 1.1 criteria [100]. Target lesions selected for tumor measurements should be those where additional (e.g., palliative) treatments are not indicated or anticipated.
* All residual toxicity related to prior anticancer therapies (excluding alopecia, grade 2 fatigue, vitiligo, endocrinopathies on stable replacement therapy, grade 2 neuropathy from taxanes or platinum and grade 2 hearing loss from platinum) must resolve to grade 1 severity or less (or returned to baseline) prior to receipt of study treatment.
* Read, understood, and provided written informed consent, and if applicable, Health Insurance Portability and Accountability Act (HIPAA) authorization, after the nature of the study has been fully explained, and must be willing to comply with all study requirements and procedures.

Exclusion Criteria:

* Among any patients enrolled in the first line treatment setting, tumors should not be PD-L1+ by 22C3 assays or eligible for FDA approved standard of care chemotherapy and anti-PD-1/PD-L1 combination therapy as alternative to this clinical trial. This does not apply if patients have previously received PD-1 or PD-L1 blockade as part of neoadjuvant or adjuvant therapy regimen.
* History of severe hypersensitivity reactions to mAbs.
* Prior treatment with any anti-CD40 antibody or rhuFlt3L product.
* Treatment with anthracycline in the metastatic setting.
* Prior progression while on anthracycline based therapy or within 6 months of completing neoadjuvant or adjuvant anthracycline.
* Prior history of acute myeloid leukemia (AML), or tumor with known Flt3 mutation/amplification
* Receipt of any antibody targeting T cell check point or co-stimulation pathways within 4 weeks, use of any other monoclonal based therapies within 4 weeks, and all other immunotherapy (tumor vaccine, cytokine, or growth factor given to control the cancer) within 2 weeks prior to the planned start of study treatment.
* Prior T-cell or other cell-based therapies within 12 weeks (or 2 weeks if patient experienced disease progression on the prior treatment)
* Systemic radiation therapy within 4 weeks, prior focal radiotherapy within 2 weeks, or radiopharmaceuticals (strontium, samarium) within 8 weeks prior to the first dose of study treatment.
* Chemotherapy or antibody drug conjugate within 21 days or at least 5 half-lives (whichever is shorter) prior to the planned start of study treatment.
* Any kinase inhibitors within 2 weeks prior to the first dose of study treatment.
* Major surgery within 4 weeks prior to the first dose of study treatment. Surgery requiring local/epidural anesthesia must be completed at least 72 hours before study drug administration and patients should be recovered.
* Use of other investigational drugs within 4 weeks or 5 half-lives (whichever is longer) prior to study treatment administration.
* Use of immunosuppressive medications within 4 weeks or systemic corticosteroids within 2 weeks prior to first dose of study treatment. Topical, inhaled or intranasal corticosteroids (with minimal systemic absorption) may be continued if the patient is on a stable dose. Non-absorbed intraarticular corticosteroid and replacement steroids (≤ 10 mg/day prednisone or equivalent) will be permitted.
* Other prior malignancy, except for adequately treated basal or squamous cell skin cancer or in situ cancers; or any other cancer from which the patient has been disease-free for at least 3 years.
* Active, untreated central nervous system metastases.
* Patients with known treated brain metastases should be neurologically stable for 4 weeks post-treatment and prior to study enrollment. Continued use of steroids and/or anticonvulsants (in the absence of any suspicion of progressive brain metastases) is acceptable if ≤ equivalent of prednisone 10 mg daily. Brain MRI required on screening to document lack of progression.
* Women who are pregnant or nursing. All female patients with reproductive potential must have a negative pregnancy test prior to starting treatment.
* Active autoimmune disease or history of autoimmune disease or syndrome that required systemic steroids or immunosuppressive medications within the preceding 6 months, except for patients with vitiligo, endocrinopathies, or type 1 diabetes, Patients with mild asthma who require intermittent use of bronchodilators (such as albuterol) who have not been hospitalized for asthma in the preceding 6 months will not be excluded from this study.
* Significant cardiovascular disease including unstable angina pectoris, uncontrolled hypertension or arrhythmia, congestive heart failure (New York Heart Association Class III or IV or EF<50%) related to primary cardiac disease, uncontrolled ischemic or severe valvular heart disease or any of the following within 6 months prior to the first dose of study treatment: myocardial infarction, severe/unstable angina, coronary artery bypass graft, congestive heart failure, cerebrovascular accident, transient ischemic attack.
* For patients with triple negative breast cancer- prior anthracycline therapy with a cumulative doxorubicin-equivalent dose greater than 240 mg/m2. 240 mg/m2 anthracycline is equivalent to 4 doses of anthracycline-based chemotherapy in the localized setting (generally 60 mg/m2 per dose). Notes from physicians demonstrating 4 prior cycles/doses of anthracycline or if less than 60 mg/m2 specifying as such to estimate the total anthracycline dose is sufficient. Exact calculation based on mg received originally is not required.
* For patients with hormone receptor positive breast cancer who have received a prior anthracycline therapy with a cumulative doxorubicin-equivalent dose exceeding 240 mg/m2 (as was part of standard-of-care regimens in the past), a cardiology evaluation is recommended to minimize potential risks of heart damage.
* Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed. The COVID-19 vaccines available in the United States are not live vaccines and are allowed if the final vaccine dose (of a regimen that requires more than 1 dose) is received at least 1 week prior to study enrollment.
* History of (non-infectious) pneumonitis or has current pneumonitis. This includes asymptomatic infiltrates on screening chest CT scan that are felt by the investigator to potentially be an inflammatory process (i.e. grade 1 pneumonitis).
* Active infection requiring systemic therapy, known HIV infection, or positive test for hepatitis B surface antigen or hepatitis C (antibody screen and if positive confirmed by RNA analysis). If positive results are not indicative of a true active or chronic infection, the patient can be enrolled after discussion with and agreement by the Investigator.
* Any other acute or chronic medical or psychiatric condition or laboratory abnormality that could increase the risk associated with trial participation or trial drug administration or could interfere with the interpretation of trial results and, in the judgment of the investigator, would make the patient inappropriate for entry into the trial.
* Evidence of acute or chronic infection on screening chest radiography.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-04-20 (Actual); Primary Completion 2026-04-20 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
Safety (tolerability) of the drug combination of CDX-1140, CDX-301 and PLD as measured by the number of participants with Dose Limiting Toxicity (DLT) | Baseline up to 12 months
  DLTs are defined as toxicities that meet pre-defined severity criteria including serious Hematologic/Non-Hematologic adverse events (AEs) and AEs at Grade 3 or above; Any ≥ grade 2 eye pain or reduction of visual acuity that does not improved to ≤ grade 1 severity within 2 weeks of initiation of topical therapy or requires systemic treatment.
  Based on National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0

SECONDARY OUTCOMES:
Anti-tumor immune response by on-treatment CD8 T cell infiltrate | After Cycle 1 (~4 weeks)
  Anti-tumor immune response will be measured by on-treatment CD8 T cell infiltrate in cells/mm^2.
Change in CD8 T cell infiltrate | Baseline, After Cycle 1 (~4 weeks)
  Change in CD8 T cell infiltrate will be measured in cells/mm^2 after cycle 1 compared to baseline.
Median Progression Free Survival by RECIST v1.1 with administration of CDX-1140, CDX-301, and PLD chemotherapy. | Baseline until date of first observed disease progression or death, assessed up to12 months
  Median Progression Free Survival measured by RECIST v1.1, defined as the time from randomization to the time of radiographic progression or death from any cause during the study, whichever occurs first.
Overall Response Rate(ORR) by RECIST v1.1 with administration of CDX-1140, CDX-301, and PLD chemotherapy. | Baseline until date of first observed objective tumor response assessed up to12 months
  Best ORR by RECIST v1.1 defined as the proportion of patients with an objective tumor response (either partial response [PR] or complete response [CR] per investigator.
Duration of Response(DoR) by RECIST v1.1 to CDX-1140, CDX-301, and PLD chemotherapy. | Date of response until progression or death from any cause, assessed up to 12 months
  Duration of response (DoR) defined as the time from the first occurrence of a documented objective tumor response to the time of radiographic progression (per investigator using RECIST v1.1) or death from any cause on study, whichever occurs first.
Clinical benefit rate (CBR) by RECIST v1.1 with administration of CDX-1140, CDX-301, and PLD chemotherapy. | 6 months
  CBR defined as percentage of patients with CR, PR, or stable disease [SD] by RECIST v1.1 at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Sangeetha Reddy, Principal Investigator — University of Texas Southwestern Medical Center
Locations (7):
- United States (7):
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - University of North Carolina, Chapel Hill, North Carolina
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Texas Oncology, P.A., Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No